CLINICAL TRIAL: NCT03353792
Title: Restoring Brain Metabolism and Function in Older Adult T1DM Patients Using an AP System
Brief Title: Using an Artificial Pancreas System in Older Adult Type 1 Diabetes Mellitus Patients
Acronym: T1DM AP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Initial difficulty with recruitment was exasperated by COVID pause of the study and then the end of funding.
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000020059; 1R01DK101984-01A1 (NIH); 1DP3DK112227-01 (NIH)
Record Dates: First submitted 2017-11-09; First posted 2017-11-27 (Actual); Results first posted 2022-10-28 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Type1 Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The design is a single-site, parallel group, randomized clinical trail. Following enrollement and CGM documentation of hypoglycemia during the 4-week run-in period, study participants are randomized to intervention and control groups.
Who Masked: Participant
Masking Description: The intervention consists of treatment with a CL/AP-enabled insulin pump/CGM combination; subjects in the control group will continue their usual diabetes care (insulin pump therapy) along with CGM recording .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- CL/AP system (Active Comparator): To improved glycemic control and strict avoidance of hypoglycemia via 8-week use of a CL/AP system (closed-loop/artificial pancreas) reverses brain metabolic adaptations in older adult T1DM patients.
  Interventions: Device: CL/AP system
- usual care (Placebo Comparator): Subjects in this control group will continue their usual diabetic care (insulin pump therapy) along with CGM recording.
  Interventions: Device: usual diabetic care

INTERVENTIONS:
Device: CL/AP system — CL/AP system enabled insulin pump/CGM combination
  Arms: CL/AP system
Device: usual diabetic care — usual diabetic care (insulin pump therapy) along with CGM recording
  Arms: usual care

SUMMARY:
To demonstrate that a new insulin pump system can prevent low glucose episodes and improve brain function in aged Type 1 diabetes mellitus subjects.

DETAILED DESCRIPTION:
The goals of this proposal are to implement a Close-Loop/Artificial Pancreas (CL/AP) system in older patients with type 1 diabetes mellitus (T1DM) in order to reverse brain metabolic adaptations and restore metabolic sensitivity, hypoglycemia awareness and appropriate hormonal counterregulatory responses (CRR). For purposes of this study we are looking to enroll aged T1DM subjects under insulin pump treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Male or female
* Age 50-75 years (at least 50% over the age of 65)
* T1DM (>20 years duration)
* C-peptide undetectable
* HbA1c of < 8%
* Insulin pump therapy
* History of frequent hypoglycemia with unawareness (defined as 2 or more episodes of severe hypoglycemia within one year requiring assistance) and 2 or more glucose values < 54 mg/dL during the week of Continuous Glucose Monitoring (CGM) (iPRO monitor, Medtronic) prior to enrollment
* BMI <27 kg/m2
* Good general health as evidenced by medical history and blood screening
* Willing to comply with all study procedures and be available for the duration of the study
* Willing to fast for a limited time period on the morning of a clamp study

Exclusion Criteria:

* Significant diabetic complications (untreated proliferative retinopathy, creatinine ≥1.5 mg/dl, urinary albumin levels 300 mg/day, autonomic neuropathy, painful peripheral neuropathy)
* Significant alcohol intake and vegetarian diet since both are known to have an impact on counterregulation and brain metabolism
* Any contraindications for MRI scanning, including presence of metallic implants or claustrophobia.
* Heavy exercise on a regular basis (i.e. marathon runners)
* Known allergic reactions to components of the study product(s)
* Treatment with another investigational drug or other intervention
* Active infection including hepatitis C, hepatitis B, HIV
* Any past or current history of alcohol or substance abuse
* Psychiatric or neurological disorders under active treatment
* Baseline hemoglobin < 10.5 g/dL in females, or < 12.5 g/dL in males. Blood donation within 30 days of the study
* History of coagulopathy or medical condition requiring long-term anticoagulant therapy (low-dose aspirin treatment is allowed)
* Co-existing cardiac, liver, and kidney disease
* Abnormal liver function tests
* Women that are on oral contraceptives, post-menopausal, pregnant (as assessed by pregnancy test that will be performed on female participants at reproductive age), or lactating.
* Any medical condition or medication that, in the opinion of the investigators, will interfere with the safe completion of the study or study outcomes

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Herzog, MD, Principal Investigator — Yale School of Medicine Department of Endocrinology
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CL/AP System | Usual Care
Started | 4 | 3
Completed | 2 | 3
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Participant Unable to Manage Device | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants that were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | CL/AP System | Usual Care | Total
Number analyzed (Participants) | 4 | 3 | 7
Age, Customized [Count of Participants; unit: Participants]
  Age Categorized: 50-59 years | 0 | 2 | 2
  Age Categorized: 60-69 years | 3 | 1 | 4
  Age Categorized: 70-79 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 3 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 3 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Brain Alternate Fuel Uptake
Description: Change in brain alternate fuel uptake under hypoglycemia was measured by assessing the percent enrichment of Glutamine 4 (Gln4). Change was measured by subtracting follow up from baseline.
  Astrocytic glutamine C4 enrichment is a measure of brain acetate metabolism (an alternate fuel to glucose). Previous studies have shown that in people who have been exposed to frequent hypoglycemic episodes, glutamine C4 enrichment increases. Therefore, we expected a reduction in Glutamine C4 percent enrichment in the follow up NMR scans in the intervention group who avoided frequent hypoglycemic episodes through the CL/AP system. In addition, there is no specific cut off value used for Glutamine C4 enrichment, rather a change or reduction was expected and noted."
Time Frame: Baseline to 8 - 10 weeks
Population: Only 2 participants (per protocol complete cases) in the intervention had data that was analyzable due to technical issues that occured with the usual care group.
Measure: Mean (Standard Deviation); unit: percent enrichment of Gln4
Arm/Group | CL/AP System | Usual Care
Number analyzed (Participants) | 2 | 0
percent enrichment of Gln4
  Baseline | 10.855 (10.642) |
  Follow Up | 7.28 (8.888) |
  Change | 3.57 (1.754) |

2. Secondary Outcome: Change in Cognitive Function: MOCA
Description: The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Time to administer the MoCA is approximately 10 minutes. The total possible score is 30 points; a score of 26 or above is considered normal. Change was calculated by subtracting follow up from baseline. https://www.parkinsons.va.gov/resources/MoCA-Instructions-English.pdf
Time Frame: Baseline to 8-10 weeks
Population: Only those that completed both assessments (did not drop out) were included in the analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CL/AP System | Usual Care
Number analyzed (Participants) | 2 | 3
units on a scale
  Baseline | 23 (0) | 27 (2)
  Follow Up | 25.5 (0.707) | 29 (0)
  Change | -2.5 (0.707) | -2 (2)

3. Secondary Outcome: Change in Cognitive Function: Trail Test A
Description: Trail making test (TMT) A is a test of visual attention and task switching. It provides information about visual search speed, speed of processing and executive function. Time is measured in seconds. The typical average time to complete the test is 29 seconds, a "deficient" performance would be >78 seconds; most people are able to complete in 90 seconds. Change was calculated by subtracting follow up from baseline.
Time Frame: Baseline to 8-10 weeks
Population: Only those that completed both assessments (did not drop out) were included in the analyses.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | CL/AP System | Usual Care
Number analyzed (Participants) | 2 | 3
seconds
  Baseline | 63 (39) | 28 (11)
  Follow Up | 34 (3) | 21 (5)
  Change | 29 (42) | 7 (16)

4. Secondary Outcome: Change in Cognitive Function: Trail Test B
Description: Trail making test (TMT) B is a test of visual attention and task switching. It provides information about visual search speed, speed of processing and executive function. Time will be measured in seconds. The typical average time to complete the test is 75 seconds, a "deficient" performance would be >273 seconds; most people are able to complete in 180 seconds. Change was calculated by subtracting follow up from baseline.
Time Frame: Baseline to 8-10 weeks
Population: Only those that completed both assessments (did not drop out) were included in the analyses.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | CL/AP System | Usual Care
Number analyzed (Participants) | 2 | 3
seconds
  Baseline | 86 (22) | 54 (13)
  Follow Up | 68 (23) | 42 (7)
  Change | 18 (1) | 12 (17)

5. Secondary Outcome: Change in Cognitive Function: Grooved Pegboard Test
Description: The grooved pegboard test is a manipulative dexterity test that assessed psychomotor speed, fine motor control, and rapid-visual motor coordination. It consists of a small board of holes with randomly positioned slots. Pegs with a key along one side must be rotated to match the hole before they can be inserted. The task was completed using the dominant hand. Time was measured in seconds.
Time Frame: Baseline to 8-10 weeks
Population: Only those that completed both assessments (did not drop out) were included in the analyses.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | CL/AP System | Usual Care
Number analyzed (Participants) | 2 | 3
seconds
  Baseline | 105 (64) | 78 (13)
  Follow Up | 100 (53) | 73 (18)
  Change | 5 (11) | 5 (8)

ADVERSE EVENTS:
Time Frame: Up to 10 weeks
Arm/Group | CL/AP System | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 0/4 | 0/3

LIMITATIONS AND CAVEATS:
This study experienced low enrollment prior to being paused due to COVID19. Upon restart of the study, it was determined that there were not sufficient funds to fully resume the trial. The overall enrollment did not provide adequate numbers to perform statistical analyses outside of providing summary statistics on those that were enrolled and those that completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/92/NCT03353792/Prot_SAP_000.pdf